CLINICAL TRIAL: NCT02756650
Title: An Open Label, Exploratory Study to Establish the Efficacy and Safety of 1 Year Canakinumab Treatment in Behçet's Disease Patients With Neurologic or Vascular Involvement
Brief Title: 1 Year of Treatment With Canakinumab in Behçet's Disease Patients With Neurologic or Vascular Involvement
Acronym: Behcet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885NTR01
Record Dates: First submitted 2016-03-31; First posted 2016-04-29 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Behcet Disease
Keywords: Behcet Disease; Inflammation; Immune system; Arthritis
MeSH Terms: conditions — Behcet Syndrome; Inflammation; Arthritis | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Canakinumab (Experimental): Canakinumab was administered monthly
  Interventions: Drug: Canakinumab

INTERVENTIONS:
Drug: Canakinumab — 150 mg or 300 mg of canakinumab was administered monthly. IV (SC after month 6)
  Other Names: ACZ885

SUMMARY:
Primary objective of the study was to evaluate the safety and efficacy of canakinumab on the clinical and inflammatory findings of Behced Disease patients with neurologic and vascular involvement.

DETAILED DESCRIPTION:
Primary endpoint: Resolution of acute exacerbation findings related to Behçet's Disease (BD) based on achievements in any of the following items without deterioration on day 30:

For patients with parenchymal neurologic disease: Resolution of acute exacerbation of parenchymal neurologic findings based on improvements in any of the following items without deterioration on Day 30:

* Improvement of muscle strength, ataxia, or other relevant neurologic findings depending on the involved region on neurological examination (by Neuro-Behçet's Disease Score, Modified Expanded Disability Status Scale, and Modified Rankin Scores) cerebrospinal fluid
* Improvement in systemic inflammatory findings (CRP, Erythrocyte Sedimentation Rate , SAA)
* Any decrease in the size of the MRI lesion, or disappearance of contrast enhancement
* Improvement in patients' and physicians global assessment using a 10-cm visual analogue scale (VAS)

Complete response was defined as full clinical recovery to the pre-attack state, disappearance of MRI lesion(s), and normalisation of Cerebrospinal Fluid findings.

Partial response was defined as partial improvement in clinical findings, but with findings still worse than the pre-attack state, and MRI lesions, which become smaller with no or less enhancement, and a decrease in cerebrospinal fluid cell count.

Non-response was defined as no improvement in clinical findings, no change on MRI, no change in cerebrospinal fluid parameters, or worsening in those findings.

For patients with large vessel vascular disease: Resolution of acute vascular exacerbation findings related to Behçet's Disease based on achievements in any of the following items without deterioration at 1 month:

* Improvement in relevant symptoms (localised pain, abdominal pain, calf thickness, haemoptysis) by using physician and patient's global assessment with VAS
* Improvement in systemic inflammatory findings (CRP, ESR, SAA)
* Any improvement in radiological findings depending on the involved vessels (MR, CT or Doppler findings)
* Improvement in patients' and physicians global assessment using a 10-cm visual analogue scale (VAS)

Complete response was defined as clinical and laboratory improvement based on ≥50% improvements in patient's and physician's global assessments by using VAS, and ≥50% reduction in CRP values; along with stable or ≥20% reduced aneurysm size in patients with arterial involvement, and stable or ≥20% reduced calf swelling in patients with lower extremity venous thrombosis.

Partial response was defined as clinical and laboratory improvement based on observations of an improvement between 20-49% according to patient's and physician's global assessments by using VAS, 20-49% reduction in CRP values; along with stable or less than 20% reduced aneurysm size in patients with arterial involvement, and stable or less than 20% reduced calf swelling in patients with lower extremity thrombosis.

Non-response will be defined as observing no or less than 20% clinical improvement by patient's and physician's global VAS or worsening of clinical findings, no change or increase in acute phase response, increase in aneurysm size for patients with arterial involvement or progression of venous thrombosis in patients with venous involvement.

ELIGIBILITY:
Inclusion Criteria:

Patients aged over 18-60 Behced Disease fulfilling the International Study Group (ISG) criteria, who have a recent exacerbation of large-vessel vascular disease and/or parenchymal neurologic disease For Neurologic Involvement

* Patients experiencing an acute exacerbation of parenchymal neurologic disease involving brainstem and/or diencephalic region.
* Exacerbation is defined based on the presence of both of the following:
* An acute/subacute neurological syndrome including any of hemiparesis, ataxia, dysarthria,headache within the first month of onset of neurologic manifestations (without any prior high dose steroid treatment)
* Compatible cranial MRI lesion involving brainstem and/or diencephalic region

For Vascular Disease :

Patients experiencing an acute exacerbation of vascular disease within the last month, involving

* Large arteries (abdominal aorta, pulmonary arteries, extremity arteries)
* Large veins (deep vein thrombosis of extremities, caval vein thrombosis, dural sinus thrombosis)
* Compatible radiological findings (spiral CT, MR, or Doppler ultrasonography)

Exclusion Criteria:

For Neurologic Involvement :

* Presence of severe neurological sequelae from any previous attacks rendering the patient dependent on others physically or mentally
* Any other neurological cause underlying the picture including ischemic central nervous system lesion on MRI
* Any previous treatment with biological agents other than interferon-alpha or any previous treatment with cyclophosphamide
* No interferon in the last 6 months, no Intra Venous Metilprednizolon in the past month

For Vascular disease and general :

* Presence of severe vascular sequelae from any previous attacks rendering the patient dependent on others
* Any other vascular disease complication the evaluation of exacerbation
* Any previous treatment with biological agents other than interferon alpha, or any previous treatment with cyclophosphamide
* No interferon alpha in the last 6 months, no IVMP in the past month
* History of Squamo Cell Carcinoma OR Basal Cell Carcinoma in previous 5 years. General
* Presence or history of any other inflammatory rheumatic disease
* Positive Purified Protein Derivative test (according to local guidance) where an active Tuberculosis infection cannot be excluded via Quantiferon (T-Spot or radiographic imaging if needed) Pregnancy or lactation
* Presence of any active or chronic infection or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 30 days or oral antibiotics within 14 days prior to screening
* History or a malignancy within the last 5 years, except for successfully excised squamous or basal cell carcinoma of the skin
* Women of childbearing potential not using the contraception method(s) specified in this study, as well as women who are breastfeeding
* With known sensitivity to canakinumab
* Use of any other investigational agent in the last 30 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Gül, Prof, Study Chair — IU Faculty of Medicine; Murat Kurtuncu, Ass.Prof, Principal Investigator — IU Faculty of Medicine; Gulsen Akman Demir, Prof, Principal Investigator — Bilim University Faculty of Medicine
Locations (1):
- Novartis Investigative Site, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The publication has been planned for Q4 2020.
Access Criteria: Access from peer reviewed journal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8 subjects enrolled 5 subjects were evaluated in Rheumatology clinic. 3 subjects were evaluated in Neurology clinic.
Pre-assignment Details: Ten patients were planned to be enrolled. Nine patients were screened. Eight patients were enrolled. Six patients completed the study. One patient was dropped out in the 7th visit because of an unknown drug abuse. One patient was dropped out in the 11th visit because of adverse event, worsening in pulmonary artery aneurysm.
Groups:
- ACZ885N: Canakinumab
Period: Overall Study
Arm/Group | ACZ885N
Started | 8
Completed | 6
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Randomized Set
Arm/Group | ACZ885N
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.25 (2.320)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Attacks
Description: Resolution of acute exacerbation findings related to Behçet's Disease (BD). The attacks were assessed by pyhsician global assesment.
  For patients with parenchymal neurologic disease: Resolution of acute exacerbation of parenchymal neurologic findings based on improvements in any of the following items without deterioration on Day 30
  This was an exploratory trial that was not powered for a statistical analysis.
Time Frame: 30 days
Population: Intent-to-Treat (ITT) population: all 8 subjects who took at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | ACZ885N
Number analyzed (Participants) | 8
Participants | 0

2. Primary Outcome: Modified Expanded Disability Status Scale (EDSS)
Description: The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with MS. Scale range is between 0-10 with 10 being most disability. Mean score of 3 participants who were evaluated in Neurology clinic. Other 5 participants were not evaluated for EDSS.
Time Frame: 30 days
Population: Behçet's Disease set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ACZ885N
Number analyzed (Participants) | 3
scores on a scale | 1.16 (2.02)

3. Primary Outcome: Neuro-Behçet's Disability Score (NBDS)
Description: Neuro-Behçet's disability score (NBDS) has been proposed for parenchymal-NBD patients to quantify disabilities. This comprises scores for motor and cognitive status. NBDS is the arithmetic sum of both scores and ranges from 0 to 8, with 8 being death due to NBD. 3 neurologic participants were evaluated.
Time Frame: 30 days
Population: Behçet's disease set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ACZ885N
Number analyzed (Participants) | 3
scores on a scale | 0.66 (1.15)

4. Primary Outcome: Modified Ranking Score (mRS)
Description: Mean Modified Rankin Scale (mRS): mRS is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Scores range from 0-5 with 5 being the worst outcome. Only 3 participants from neurology clinic were evaluated with this scale.
Time Frame: 30 days
Population: Behçet's disease set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ACZ885N
Number analyzed (Participants) | 3
scores on a scale | 0.66 (1.15)

5. Primary Outcome: Ataxia
Description: Number of the partcipants with ataxia. 3 participants from neurology clinic were evaluated.
Time Frame: 30 days
Population: Randomized set
Measure: Count of Participants; unit: Participants
Arm/Group | ACZ885N
Number analyzed (Participants) | 3
Participants | 1

6. Primary Outcome: Physical Examination Scores Indicating Change in Muscle Strength
Description: All 4 extremties were evaluated for muscle strength (upper right, upper left, lower right and lower left) fro each patient. Score 0 is the worst outcome whereas 5 is the best outcome for muscle strength. 3 participants from neurology clinic were assessed.
Time Frame: 30 days
Population: Behçet's disease set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ACZ885N
Number analyzed (Participants) | 3
scores on a scale
  Upper right extremity | 5.0 (0)
  Lower right extremity | 5.0 (0)
  Upper left extremity | 4.7 (0.57)
  Lower left extremity | 5.0 (0)

7. Primary Outcome: C-reactive Protein (CRP) Values
Description: Mean CRP (C-reactive protein) value (8 participants)
Time Frame: 30 days
Population: randomized set
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ACZ885N
Number analyzed (Participants) | 8
mg/L | 14.58 (20.26)

8. Primary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: Mean erythrocyte sedimentation rate (ESR) value (8 participants)
Time Frame: 30 days
Population: randomized set
Measure: Mean (Standard Deviation); unit: mm/H
Arm/Group | ACZ885N
Number analyzed (Participants) | 8
mm/H | 17.5 (12.77)

9. Primary Outcome: SAA (Serum Amyloid A)
Description: Mean Serum Amyloid A value (8 participants)
Time Frame: 30 days
Population: randomized set
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ACZ885N
Number analyzed (Participants) | 8
mg/L | 78.66 (108.17)

10. Primary Outcome: Hemoptysis
Description: The number of the participants with hemoptysis
Time Frame: 30 days
Population: randomized set
Measure: Count of Participants; unit: Participants
Arm/Group | ACZ885N
Number analyzed (Participants) | 8
Participants | 1

11. Primary Outcome: Visual Analogue Scores (VAS) for Headache
Description: Headache intensity was measured by VAS where score 0 means "no pain," and score 10 means "the worst pain''. Physician and participant determined the VAS score separately.
Time Frame: 30 days
Population: randomized set
Measure: Mean (Standard Deviation); unit: average of scores on a scale
Arm/Group | ACZ885N
Number analyzed (Participants) | 8
average of scores on a scale
  VAS by participants | 0.27 (0.32)
  VAS by Physicians | 0.2 (0.18)

12. Primary Outcome: Visual Analogue Scores (VAS) for Stomachache
Description: Stomacheache intensity was measured by VAS where score 0 means "no pain," and score 10 means "the worst pain''. VAS is determined separately by physician and the participants.
Time Frame: 30 days
Population: randomized set
Measure: Mean (Standard Deviation); unit: average of scores on a scale
Arm/Group | ACZ885N
Number analyzed (Participants) | 8
average of scores on a scale
  VAS by participants | 0.27 (0.32)
  VAS by physicians | 0.18 (0.17)

13. Primary Outcome: Visual Analogue Scores (VAS) for Extremity Assessments
Description: Extremity assessments were measured by VAS where score 0 means "no pain," and score 10 means "the worst possible pain''. The physicians and participants evaluated VAS separately.
Time Frame: 30 days
Population: randomized set
Measure: Mean (Standard Deviation); unit: average of scores on a scale
Arm/Group | ACZ885N
Number analyzed (Participants) | 8
average of scores on a scale
  VAS by participants | 1.07 (1.13)
  VAS by physicians | 0.87 (0.98)

14. Primary Outcome: Visual Analogue Scores (VAS) for Patients' General Assessments
Description: Participants assessed their own well-being with VAS (visual analogue scale). Score 0 means the best outcome, score 10 is the worst outcome.
Time Frame: 30 days
Population: randomized set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ACZ885N
Number analyzed (Participants) | 8
scores on a scale | 1.72 (1.36)

15. Primary Outcome: Physician's Global Assessment
Description: Physician's General Assessments is VAS scale, ranging between 0-5, showing the disease status of participants. Score 0 is the worst outcome; 5 is the best outcome
Time Frame: 30 days
Population: randomized set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ACZ885N
Number analyzed (Participants) | 8
scores on a scale | 3.75 (0.46)

16. Primary Outcome: Steroid Dose Regimen
Description: Mean steroid treatment dose (8 participants)
Time Frame: 30 days
Population: randomized set
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | ACZ885N
Number analyzed (Participants) | 8
mg/day | 9.5 (2.73)

17. Primary Outcome: BDCAF (Behçet's Disease Current Activity Form)
Description: BDCAF is an assessment that is made by physician for evaluating the disease activity in last four weeks. Score range is 0 to 12, 0 is the best outcome, 12 is the worst outcome.
Time Frame: 30 days
Population: randomized set
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | ACZ885N
Number analyzed (Participants) | 8
scores | 1.62 (1.5)

18. Primary Outcome: Extremity (Localized) Pain Assessment (VAS)
Description: Localized pain in the extremities were assessed by visual analogue scale scores ranging between Scale; 0 is the best outcome; 10 is worst.
Time Frame: 30 days
Population: randomized set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ACZ885N
Number analyzed (Participants) | 8
scores on a scale | 1.28 (1.22)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment
Description: An AE is any sign or symptom that occurs during the study treatment plus the # days post treatment
Arm/Group | ACZ885N
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885N (N=8)
Middle ear inflammation (Ear and labyrinth disorders) | 1
Swelling of eyelid (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Aphthous ulcer (Gastrointestinal disorders) | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Folliculitis (Infections and infestations) | 3
Influenza (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Nystagmus (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Genital ulceration (Reproductive system and breast disorders) | 1
Testicular swelling (Reproductive system and breast disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary artery aneurysm (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 2
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
This was an exploratory trial that was not powered for a statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT02756650/Prot_SAP_000.pdf